CLINICAL TRIAL: NCT06951737
Title: Evaluation Of The Effect Of SGLT-2 Inhibitors On Atrial Fibrillation Recurrence In Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Bursa Postgraduate Hospital (Other)
Responsible Party: Principal Investigator, Hasan ARI, Prof Dr, Bursa Postgraduate Hospital
Other Study IDs: Bursa SUAM
Record Dates: First submitted 2025-04-20; First posted 2025-04-30 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus; Atrial Fibrillation (AF)
MeSH Terms: conditions — Diabetes Mellitus; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SGLT-2 inhibitor user: patients with diabetes mellitus, atrial fibrillation and using SGLT-2 inhibitor

SUMMARY:
Consecutive DCCV was performed until to achieve 120 patients in SR (60 DM patients who used SGLT-2 inhibitors and 60 DM patients who did not use SGLT-2 inhibitors). Patients defined as SGLT-2 inhibitor user group and control group. The two groups were monitored for AF recurrence on the first day, then at one, three, and six months after CV.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years and < 90 years,
* Patient diagnosed with DM
* Patient underwent electrical cardioversion due to AF and was restored to sinus rhythm

Exclusion Criteria:

* patient who are not suitable for anticoagulant use,
* have thyroid dysfunction,
* glomerular filtration rate ≤ 25 ml/min/1.73 m²,
* patients whose sinus rhythm cannot be achieved with electrical cardioversion,
* malignancy patients,
* patients with acute or chronic inflammatory disease,
* patients with peripheral artery disease,
* patients with pacemakers,
* patients with advanced valve stenosis or insufficiency,
* patients who have had coronary bypass surgery,
* patients with percutaneous or surgical bioprosthesis or metallic valve surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with DM and AF who were planned to undergo electrical cardioversion were evaluated for suitability for the study.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-10-02 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence | six month

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yüksek İhtisas Hastanesi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yarar M, Ari H, Ari S, Tutuncu A, Melek M, Bozat T. Evaluation of the effect of SGLT-2 inhibitors on atrial fibrillation recurrence in diabetic patients. Expert Opin Pharmacother. 2025 Aug;26(11-12):1343-1349. doi: 10.1080/14656566.2025.2527189. Epub 2025 Jul 3. PMID 40579747